CLINICAL TRIAL: NCT04138433
Title: Mechanisms Underlying Spoken Language Production: Facilitating Frontal Brain Networks Following Aphasic Stroke
Brief Title: Mechanisms Underlying Spoken Language Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Jenny Crinion, Professor Jennifer Crinion, University College, London
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 160106
Record Dates: First submitted 2016-10-24; First posted 2019-10-24 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aphasia, Anomic
MeSH Terms: conditions — Anomia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): fMRI task plus anodal tDCS
  Interventions: Device: Real tDCS
- Sham tDCS (Sham Comparator): fMRI task plus sham tDCS
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Real tDCS — Anodal tDCS 2 ma
  Other Names: Brain Stimulation
  Arms: Real tDCS
Device: Sham tDCS — Sham tDCS 2 ma
  Other Names: Brain Stimulation
  Arms: Sham tDCS

SUMMARY:
Most of us take being able to communicate for granted. Anomia (word finding problems) after stroke can cause profound frustration and anxiety for patients and families. Some people recover; many don't. ~ 250,000 people in the UK have chronic speech and language problems post-stroke. This project will investigate how treatment for these people might be improved. The brain's speech areas can be stimulated using transcranial direct current stimulation (tDCS). The kit is simple; a battery powering electrodes placed on the scalp. Healthy people who had tDCS while naming pictures could find words quicker and their speech areas responded more efficiently. How it affects aphasic stroke patients' brain function is unknown.

DETAILED DESCRIPTION:
All suitable participants will be living in the community and may have already consented to previous research projects and their details identified via the UCLH Aphasia Clinic run by the CI, which will act as an NHS PIC, or via the stroke volunteer database at the Wellcome Trust Centre for Neuroimaging, run by Professor Cathy Price (Research approved by the National Hospital of Neurology and Neurosurgery and the Institute of Neurology joint ethics committee, study number: NO32.

The initial approach to potential participants for this project will be made by The Chief Investigator Dr Jenny Crinion. If the participant agrees a member of the team will discuss with them the details of the project. Patient groups may be approached directly by the CI and RAs via stroke clubs etc. All participants will be formally consented at UCL.

Healthy subjects will be recruited by the CI and RAs via the volunteer database at the WTCN or ICN, and by asking relatives/carers of the patients if they wish to be involved (more likely to be matched for age and other factors). Potential participants in research databases have already consented to be approached for further research.

Part 1: Activation and modulation of residual inferior frontal gyrus (IFG) in aphasia

Aims: to examine connectivity within regions of the brain associated with spoken word retrieval (a "domain-specific" process) and more general cognitive control ("domain-general" processing) in aphasic stroke patients.

Hypotheses: following aphasic stroke a functionally selective network core for spoken word naming (i.e. domain specific for language) lies within (i) Broca's area, in patients with brain lesions sparing Broca's area (ii) right inferior frontal gyrus, in patients with damage to Broca's area.

Experimental design and predictions:

Patients with a chronic speech and language impairment (aphasia) following stroke will be divided into those with lesions affecting Broca's area, and those whose lesions lie elsewhere. They will receive brain stimulation, transcranial direct current stimulation (tDCS, which involves placing battery-operated electrodes on the participant's scalp), or sham stimulation, while completing an object naming task (to test domain-specific processing) and a non-linguistic task which measures performance related to domain-general cognitive processing. Both tasks will have "hard" and "easy" levels which are matched for difficulty across tasks. In the naming task, difficulty will be manipulated by providing different types of cues to assist with object naming. Extensive piloting of the stimuli and procedure in both healthy participants and aphasic stroke patients will ensure that the tests are suitable for the proposed research.

Participants will complete the experiment in an MRI scanner in order to measure brain activity in the domain-specific and domain-general neural networks during the linguistic and non-linguistic tasks.

List of all data to be collected

1. Personal demographic data including: sex, age, contact details etc.
2. Clinical data including: aphasic syndrome subtype, time since onset of symptoms, past medical history, current medications, contra-indications to MRI/fMRI/tDCS, etc.
3. Language assessment scores (CAT).
4. Naming scores.
5. fMRI responses when speaking and at rest.
6. High-resolution structural MRI scans to define area and volume of infarct
7. Side-effects from stimulation/sham (Adverse Event data).
8. Consent forms. The non-functional imaging data will be recorded on a Case Report Form (CRF) kept by the CI.

Collection/Storage

Any data initially collected on paper will be transferred to electronic format. The paper data (including a copy of the consent form) is stored in a locked cabinet at the ICN which only the CI and named collaborators will have access to. The electronic data is password protected and pseudoanonymized. The CI will be the custodian of the data after the trial is completed. Data will be kept for 10 years after the completion of the study, in line with UCL policy. The functional/structural imaging data (5, 6) will be stored indefinitely at the WTCN, this will be password protected. These are extremely rich data sets and may be used in future analyses/metanalyses. Only members of the research team will have access to the data. The CI will act as custodian of the data.

Monitoring and Auditing

The Chief Investigator will ensure there are adequate quality and number of monitoring activities conducted by the study team. This will include adherence to the protocol, procedures for consenting and ensure adequate data quality. The Chief Investigator will inform the sponsor should he/she have concerns which have arisen from monitoring activities, and/or if there are problems with oversight/monitoring procedures. An independent data monitoring committee (DMC) will be set up to deal with patient safety issues related to this project.

The data to be monitored by the DMC will include: language outcome scores (CAT) and Adverse Event Recording Forms. All adverse events will be recorded by the CI and passed on to the DMC and will follow the UCL protocol for reporting of adverse events in a single centre trial. The main function of the committee will be to determine if there is an excess of seizures (adverse events) in either patient group. There are no plans to stop the project early unless this is due to an excess of adverse events.

ELIGIBILITY:
* Inclusion criteria, subjects will be:

  1. English native speakers
  2. Over the age of 18
  3. 12 months or more after aphasic stroke
  4. Able to provide informed consent
* Exclusion criteria, subjects will not have:

  1. Significant medical or psychiatric co-morbidity
  2. Clinical or neuroimaging evidence of significant multifocal cerebral disease
  3. Contraindications to tdcs
  4. Contraindications to MRI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Naming Speed | change from baseline to 20 minutes during and 20 minutes post tDCS intervention
  change in Tailor-made object naming test,

SECONDARY OUTCOMES:
Higher accuracy in naming | change from baseline to 20 minutes during and 20 minutes post tDCS intervention
  change in scores from tailor-made object naming tests

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crinion, Dr, Principal Investigator — University College, London
Locations (1):
- Institute of Cognitive Neuroscience, University College London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No